CLINICAL TRIAL: NCT05583305
Title: Prevalence and Etiologies of Intracranial Stenosis in Patients With Antiphospholipid Syndrome: a Cross Sectional Study (ICAS_APS)
Brief Title: Prevalence and Etiologies of Intracranial Stenosis in Patients With Antiphospholipid Syndrome
Acronym: ICAS_APS
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CREC 2022.352
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Antiphospholipid Syndrome; Stenosis; Intracranial Stenosis
MeSH Terms: conditions — Antiphospholipid Syndrome; Constriction, Pathologic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with APS: Investigators shall recruit patients with the following criteria:
  1. Diagnosed with APS who fulfilled the modified Sapporo criteria:
     1. at least one clinical criterion (vascular thrombosis or pregnancy morbidity); and
     2. laboratory criteria (aPL positivity twice, 12 weeks apart):
     i. Lupus anticoagulant positivity requires screening, mixing, and confirmation test as per International Society of Thrombosis and Hemostasis guidelines (11).
     ii. Anticardiolipin antibodies positivity requires a medium to high titer IgG and/or IgM level by ELISA assays.
     iii. Anti-β2 glycoprotein antibodies positivity requires a >99th titer IgG and/or IgM level by ELISA assays.
  2. Patients age ≥18 years
  3. Patients who are able to provide an informed consent to study procedures
  Interventions: Diagnostic Test: Imaging assessment; Diagnostic Test: Neurosonology assessment; Diagnostic Test: Blood Test
- Controls: From the ongoing prospective Brain Health Longitudinal study which contained stroke- and dementia free participants (CREC Ref. No: 2018.148), investigators shall identify age- and gender-matched individuals without aPLs as controls
  Interventions: Diagnostic Test: Imaging assessment; Diagnostic Test: Neurosonology assessment; Diagnostic Test: Blood Test

INTERVENTIONS:
Diagnostic Test: Imaging assessment — Investigators shall perform cranial MRI examinations. The scanning protocol will employ an MRI scan protocol with T1-weighted, T2-weighted, FLAIR, susceptibility weighted imaging, diffusion weighted imaging, and time-of-flight magnetic resonance angiography (MRA) sequences. In addition, high-resolution magnetic resonance vessel wall imaging (HRMRI) allows assessment of the vessel wall using specific the SPACE sequence and the MATCH sequence. Assessors of the HRMRI images shall be blinded to the group allocation and clinical information.
Diagnostic Test: Neurosonology assessment — Investigators shall perform carotid duplex ultrasonography (CD) assessment, focusing on the peak systolic (PSV) and end diastolic velocity (EDV) of bilateral extracranial internal carotid arteries (ICA) Brightness mode imaging shall gauge the intimal thickness and plaque characteristics (if any) of bilateral ICAs.
Diagnostic Test: Blood Test — Nine milliliters of EDTA blood will be drawn during the research clinic visit for evaluation of the degree of neurovascular inflammation. Serum plasminogen activator inhibitor-1 (PAI-1) and high-sensitive C-reactive protein (hsCRP) are markers of vascular inflammation, atherosclerosis, and thrombotic risk. Serum neurofilament light chain (NfL) is a biomarker for neuroaxonal injury that correlates with small vessel disease.

SUMMARY:
Antiphospholipid syndrome (APS) is an important cause of young stroke which could result in major disability. Cohort studies suggested that 17% of young ischemic stroke were accountable by APS (1). Although warfarin has been the mainstay of treatment in APS for the past decades, recurrent thromboembolism occurred up to 10% of warfarinized patients with APS (2, 3). These observations call for an in-depth understanding of disease mechanisms secondary to antiphospholipid antibodies (aPL). Contrary to traditional understanding, recent evidence suggested mechanisms of cerebrovascular ischemia in APS are far more complex than hypercoagulability alone.

In the proposed cross-sectional study, we aim to determine the prevalence of intracranial stenosis, and to explore the correlations between the neuroimaging findings and the immunological as well as clinical features in patients with APS.

In the proposed cross-sectional study, we aim to determine the prevalence of intracranial stenosis, and to explore the correlations between the neuroimaging findings and the immunological as well as clinical features in patients with APS.

DETAILED DESCRIPTION:
In the proposed cross-sectional study, we aim to determine the prevalence of intracranial stenosis, and to explore the correlations between the neuroimaging findings and the immunological as well as clinical features in patients with APS.

Upon reviewing the clinical and laboratory information in the medical specialist out-patient clinics, electronic patient record and/or through the Clinical Data Analysis And Reporting System (CDARS), investigators shall identify and recruit on-site APS patients who fulfilled the modified Sapporo criteria, currently aged ≥18 years, and receive care from the Prince of Wales Hospital.

Investigators shall then arrange a study clinic visit for eligible patients. After obtaining an informed consent, patients will be subjected to cognitive assessment (Hong Kong Version of Montreal Cognitive Assessment (HK-MoCA)), blood pressure, pulse, body mass index measurement, urinalysis, and contrast MRI brain (see imaging assessment below). Demographic data (age, gender, smoking, drinking, ambulatory status), medical comorbidities (concurrent autoimmune diseases and their organ involvement, history of catastrophic APS, hypertension, hyperlipidemia, diabetes mellitus, congestive heart failure, number and type of previous arterial or venous thromboembolism), laboratory parameters (complete blood count, liver and renal function test, C-reactive protein, erythrocyte sediment rate, high sensitive C-reaction protein, plasminogen activator inhibitor-1, neurofilament light chain, titers of autoimmune markers including anti-nuclear antibodies, extractable nuclear antigen antibodies, aPLs, rheumatoid factor, anti-cyclic citrullinated peptide antibody, etc.), concurrent medications (aspirin, warfarin, direct oral anticoagulants, antihypertensives, statins, steroid, immunosuppressants, etc.). In another ongoing prospective Brain Health Longitudinal study which contained stroke- and dementia free participants (CREC Ref. No: 2018.148), investigators shall identify age- and gender-matched individuals without aPLs as controls. They will be assessed in the same manner as the APS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with APS who fulfilled the modified Sapporo criteria:

   1. at least one clinical criterion (vascular thrombosis or pregnancy morbidity); and
   2. laboratory criteria (aPL positivity twice, 12 weeks apart):

   i. Lupus anticoagulant positivity requires screening, mixing, and confirmation test as per International Society of Thrombosis and Hemostasis guidelines (11). ii. Anticardiolipin antibodies positivity requires a medium to high titer IgG and/or IgM level by ELISA assays. iii. Anti-β2 glycoprotein antibodies positivity requires a >99th titer IgG and/or IgM level by ELISA assays.
2. Patients age ≥18 years
3. Patients who are able to provide an informed consent to study procedures

Exclusion Criteria:

1. Patient with established neurological disease, such as stroke, cerebral venous thrombosis, vasculitis of the central nervous system, cerebral lupus, etc.
2. Patient contraindicated to contrast MRI scans. E.g. claustrophobia, allergy to gadolinium contrast, MRI incompatible implants, estimated glomerular filtration rate of < 30mL/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with or without APS
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Radiological evidence of intracranial arterial stenosis | 31／01／2026
  Defined as the presence of >50% stenosis of any intracranial arteries (ICA, MCA, anterior cerebral arteries, posterior cerebral arteries, basilar artery, or vertebral arteries) or presence of arterial plaques in vessel wall imaging.

SECONDARY OUTCOMES:
Other radiological outcomes | 31／01／2026
  Including the presence and pattern of enhancing intracranial plaques (concentric vs eccentric), Age-related White Matter Change Scale ≥ 2, white matter hyperintensity volume, presence of lacunes, cerebral microbleeds, extracranial ICA plaques, normalized total brain volume. Secondary biochemical outcomes include level of hs-CRP and PAI-1. The relationship between the neuroimaging outcomes and the clinical characteristics of patients with APS will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming IP, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No